CLINICAL TRIAL: NCT03185052
Title: Feasibility of Outpatient Care After Manual Compression in Patients Treated for Peripheral Arterial Disease by Endovascular Technique With 5F Sheath Femoral Approach
Acronym: FREEDOM OP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RC16_0384
Record Dates: First submitted 2017-06-07; First posted 2017-06-14 (Actual); Last update posted 2019-11-21 (Actual); Status verified 2019-11

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Manual puncture point compression (Other): Manual puncture point compression following a diagnostic or therapeutic procedure by endovascular technique involving retrograde femoral puncture point with 5F guide catheter
  Interventions: Other: Manual puncture point compression

INTERVENTIONS:
Other: Manual puncture point compression — Manual puncture point compression following a diagnostic or therapeutic procedure by endovascular technique involving retrograde femoral puncture point with 5F guide catheter

SUMMARY:
Over the past years, arterial closure systems have tended to replace manual compression to ensure hemostasis at femoral artery puncture points. Arterial closure systems reduce hemostasis and patient immobilization times, thus enabling early resumption of walking. These devices have contributed extensively to the development of outpatient stays for cardiology, vascular and neuro-radiology procedures.

According to certain studies however, it would appear that arterial closure devices do not present any greater benefits than manual compression in terms of hemostasis and complications. Moreover, the use of increasingly small diameter instruments would tend to render manual compression sufficient. Finally, the use of these devices generates additional costs.

The purpose of our prospective study is to evaluate the feasibility and safety of same-day discharge after manual compression in patients treated for peripheral artery disease by endovascular technique with 5F sheath.

DETAILED DESCRIPTION:
The reference management strategies for patients treated for peripheral arterial disease by endovascular technique are conventional hospitalization with manual compression and discharge after at least one over-night observation and outpatient hospitalization with the use of an arterial closure device. There are currently no official guidelines for guiding the patient towards one or other of these types of care. Indeed, outpatient management of artery disease is implemented in only a few centers in France. Several studies have shown that outpatient care is perfectly safe for patients. Our experiment at the Nantes University Hospital demonstrates also the reliability and safety of this care through the use of closure systems as shown by Albert. Now, it seems judicious to develop and improve this care since the use of smaller diameter devices would tend to render manual compression sufficient.

The method used is based on our previous protocols, routine practice and evaluation. First of all, patients eligible for same-day discharge are first selected according to SFAR (Société Française d'Anesthésie Réanimation - French Society for Anesthesia and Resuscitation) criteria for outpatients. Patients failing to meet these criteria are directed towards conventional hospitalization.

For outpatients, the patients are hospitalized in a specific unit hosting outpatients of different medico-surgical specialties. The paramedical team checks the prerequisites and the preoperative assessment. The use of a common femoral approach with 5F sheath is required. According to patients' needs, femoral anterograde or retrograde puncture are performed under duplex scan guidance. Aortoiliac and infrainguinal occlusive lesions are indifferently treated but the endovascular treatment must be compatible with the use of a stent or a drug coating balloon 5F sheath and 0.035 compatible..

The procedure should be finished 5h prior the outpatients unit closing to allow 5h follow-up. The intervention proceeded after an intravenous bolus of heparin. Anesthesia, antiplatelet regimen were let at the discretion of the interventionnalist. End-of-procedure hemostasis shall be implemented by the operator by manual compression for at least 10 minutes, potentially extended until complete hemostasis is achieved. A pressure pad shall be applied just after the end of manual compression.

The patient's general and local condition shall be monitored in the recovery room. If there are no local or general complications, the patient shall return to the ambulatory unit. In the unit, at H4, the compressive dressing is removed, patient is place in half-sitting position and without any complications, the ability to be discharged will be evaluated. The day after the operation, the patient is contacted by the ambulatory unit according with HAS and SFAR recommandations for a medical checkpoint. All of this will be conducted under medical and paramedical supervision. In the event of femoral puncture site active bleeding at any stage during care, the patient's surgeon will be notified and an additional manual compression will be applied if necessary. There are no specific guidelines concerning treatment with platelet aggregation inhibitors, whose choice will be left to the operator's discretion. In all cases, the treatments will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years,
* Endovascular treatment by stent or drug coating balloon 5F and 0.035 compatible
* Femoral approach
* Outpatient hospitalization
* Manual compression at puncture site
* Rutherford 2 to 5
* Patient affiliated with a social security scheme
* Patient's signed informed consent form

Exclusion Criteria:

* Under-age patient
* Patient of age, but under legal guardianship or care
* Contraindication to endovascular treatment
* Use of a 6F or greater sheath
* Radial or brachial puncture
* Acute ischemia
* Anticoagulant treatment or hemostasis disorder
* Allergy to Elastoplast® type adhesive strips
* Life expectancy of less than one month
* Refusal of patient to participate in the study
* Participation in another therapeutic trial
* Pregnant woman, lactating women
* Patients do not understand the French language or unfit for proposed follow in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2017-09-27 (Actual); Primary Completion 2019-10-10 (Actual); Study Completion 2019-10-10 (Actual)

PRIMARY OUTCOMES:
Total in-hospital admission rate | 1 month
  Total in-hospital admission rate includes unplanned overnight surveillance and re-hospitalization rate at 1 month.

SECONDARY OUTCOMES:
Death (all causes) at 1 month. | 1 month
Unplanned overnight surveillance rate | 1 month
Re-hospitalization after discharge during M1 | 1 month
Occurrence of major events during the perioperative period (H0 to M1) | 1 month
  Occurrence of major events during the perioperative period (H0 to M1) (MACE: Major Adverse Cardiovascular Event, MALE: Major Adverse Limb Event)
Occurrence of major punctured femoral artery events during the perioperative period (H0 to M1) | 1 month
  Occurrence of major punctured femoral artery events during the perioperative period (H0 to M1), requiring prolongation of hospitalization, repeat hospitalization or repeat surgery (hematoma, hemorrhage, false aneurysm, arterio-venous fistula, infection…).
Occurrence of minor punctured femoral artery events during the perioperative period (H0 to M1), not requiring prolongation of hospitalization, repeat hospitalization or repeat surgery | 1 month
Technical success which is defined successful vascular access and completion of the endovascular procedure and immediate morphological success with less than 30% residual diameter reduction of the treated lesion on completion angiography. | 1 month
Time for groin compression and dressing. | 1 month
Freedom from target lesion revascularization (TLR) at 1 month. | 1 month
  TLR expresses the frequency of the need for repeated procedures (endovascular or surgical) due to a problem arising from the treated lesion in surviving patients with preserved limb.
Freedom from target extremity revascularization (TER) at 1 month. TER is defined as any repeat percutaneous intervention or surgical bypass of any segment of the target limb in surviving patients with preserved limb. | 1 month
Clinical success at 1 month. | 1 month
  Clinical success is defined by defined as a sustained upward shift of 1 category of the Rutherford classification for claudicants and by wound healing and rest pain resolution for patients in CLI, without the need for repeated TLR in surviving patients.
Haemodynamic improvement: of ABI-values with 0.10 as compared to baseline values or to ABI inferior or egal 0.9 at 1-month without need for repeated TLR in surviving patients. | 1 month
Quality of life evaluation (EQ5D-3L) at 1 month. | 1 month
Economic analysis endpoints | 1 month
  Resources consumed will be recorded from the intervention to one month post-operatively. We will collect hospital resources consumed (length of procedures, operative room staff, medical device used in case of manual compression's failure, hospitalizations due to complications…) and office-based care resources (medical and paramedical consultations, caregivers).

CONTACTS AND LOCATIONS:
Locations (10):
- France (10):
  - CHU de Besançon, Besançon
  - CHU de Bordeaux, Bordeaux
  - AP-HP, Hôpital Ambroise Paré, Boulogne-Billancourt
  - CHU de Clermont Ferrand, Clermont-Ferrand
  - CHU de DIJON, Dijon
  - Clinique de Fontaine-Les- Dijon, Dijon
  - Nantes University Hospital, Nantes
  - AP-HP, Hôpital Européen Georges Pompidou, Paris
  - Institut Mutualiste Montsouris, Paris
  - Clinique de l'Europe, Rouen

IPD SHARING:
Plan to Share IPD: No